CLINICAL TRIAL: NCT05264467
Title: Use of Leukocyte and and Platelet-rich Fibrin Plasma (L-PRF) for the Prevention of Anastomotic Leakage in Colorectal Anastomosis
Brief Title: Leukocyte and and Platelet-rich Fibrin Plasma for the Prevention of Anastomotic Leakage in Colorectal Anastomosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, José Vivanco Aguilar, physician, Universidad de Concepcion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UdeConcepcion
Record Dates: First submitted 2022-01-28; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Anastomotic Leak; Platelet-Rich Fibrin; Colorectal Surgery
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: A randomized one blinded experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- PRF (Experimental)
  Interventions: Biological: Platelet rich fibrin on colorectal anastomosis

INTERVENTIONS:
Biological: Platelet rich fibrin on colorectal anastomosis — Platelet rich fibrin on colorectal anastomosis
  Other Names: Control
  Arms: PRF

SUMMARY:
Anastomotic leak rate in colorectal surgery is estimated between 4 and 20 percent. Leukocyte and and platelet-rich fibrin plasma (L-PRF) is second generation platelet concentrate whose application in colorectal anastomosis in animals has shown promising results that suppose a lower leakage rate. The objective of this study was to assess the feasibility of using L-PRF in colorectal surgery and to determine the incidence of anastomotic leakage after colorectal anastomosis.

DETAILED DESCRIPTION:
Anastomotic leakage is an important and probably the most feared complication in colorectal surgery, due its high rate of morbidity, prolonged hospitalization and mortality.

The incidence of colorectal anastomotic leakage varies between 4 and 20%, and it definition is dissimilar depending on the articles reviewed. However, results from the Dutch Colorectal Surgery Audit, published in 2010 showed a global leakage rate of 11%.

To decrease this surgical complication several strategies and devices have been developed with discouraging results. Based on the scar theory of platelet concentrates, the use of platelet-rich plasma (PRF) and leukocyte and platelet-rich fibrin plasma (L-PRF) has been proposed to stimulate and improve cicatrization in colorectal anastomosis, showing promising results in animal studies.

L-PRF is a second generation platelet concentrate of better quality and simpler confection, that is obtained by a similar technique developed in France by Choukroun et al, in the absence of anticoagulants or gelling agents. Platelet concentrates and specially L- PRF are use in various areas of odontology and medicine, including colorectal surgery.

The main objective of this study was to evaluate the feasibility of using L-PRF in colorectal surgery and to determine its effect on anastomotic leakage after colorectal anastomosis.

This study was approved by the Ethical and Scientific Committee of Health Service of Concepción city (Code: 17-07-40). All participants were explained their rights and were asked for their consent to enroll them in the study. On the other hand, anonymity and confidentiality of the participants was assured during the study, as the patients personal information was not included in the research database, which was administered only by the main investigator and the statistical analyst.

This study was held following the recommendations of Helsinski Declaration and World Medical Association.

ELIGIBILITY:
Inclusion Criteria:

* Patients were submitted to elective colorectal anastomosis with mechanic anastomosis on or under the peritoneal reflection.
* Postoperative evaluation using contrast enema to objectify subclinical dehiscence.

Exclusion Criteria:

* Age under 15 years
* American Association of Anesthesiologists (ASA) grade IV or higher.
* Clinical signs of peritonitis
* Other major surgeries within 30 days of the procedure.
* Deficient nutritional state (defined by plasmatic albumin levels lower tan 2.8 mg/dl) Active treatment with corticoids and the impossibility of having contrast enema post-surgery.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Determine the incidence of anastomotic leakage after colorectal anastomosis | 30 days
  Anastomotic leak description in both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Concepción, Concepción, Chile

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05264467/Prot_SAP_000.pdf